CLINICAL TRIAL: NCT00194597
Title: Trial of Viagra' in Men With Chronic Pelvic Pain Syndrome Type III
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Illness of PI forced termination.
Sponsor: University of Washington (Other)
Collaborators: Berger, Richard E., M.D. (Individual)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 03-9558-D 02
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2008-10-22 (Estimated); Status verified 2008-10

CONDITIONS: Prostatitis
Keywords: Prostatitis
MeSH Terms: conditions — Prostatitis | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Viagra (sildenafil citrate)

SUMMARY:
Viagra is a potent 5-PDE inhibitor that causes vasodilation in the penis and, therefore, erection in men with erectile dysfunction. Our hypothesis is that Viagra may improve the symptoms of men with Chronic Pelvic Pain Syndrome based on the following assumptions:

Chronic Pelvic Pelvic Syndrome and Interstitial Cystitis involve poorly understood central and peripheral pain sensitization such as are seen in Chronic Sympathetic Dystrophy, also called Chronic Regional Pain Syndrome. This pain may be caused by constricted blood vessels resulting from past stress, injury or trauma

Viagra will dilate sympathetically constricted vessels and improve pelvic blood flow in the same manner it does in men with erectile dysfunction.

Since men with Chronic Pelvic Pain Syndrome often complain of sexual dysfunction; improving sexual function and, therefore, quality of life may improve overall well being and perception of pain.

DETAILED DESCRIPTION:
Screening Visit (Visit 1):

Patient will review and sign the study consent form. They will then be asked to complete study questionnaires regarding demographics, medical history, pelvic pain and psychological issues.

Urine will be collected and cultured for bacteria, gonorrhea and chlamydia . It will also be analyzed for white blood cells, NO and chemistry.

There will be a physical exam and prostate massage. During the prostate massage, expressed prostatic secretions will be collected and sent to the Male Fertility Lab for analysis.

Finally, he will be asked to go to the Male Fertility Lab to provide a semen sample.

Randomization:

After the subject's urine culture results have been reviewed (patient must be free of urinary tract infection to be in study), the Investigational Pharmacy will be asked to randomize the patient.

Pharmacy will then mail the patient's first month's study medication to him. He will also be mailed medication/voiding and pain diaries to fill out over the next month.

1. Month Visit (Visit 2):

   The subject will return to the Urology Clinic about 1 month after his Screening Visit (Visit 1). He will first fill out follow-up forms.

   Next, his previous month's empty medication container and completed diaries will be collected. A pill count will then be done

   Finally, the subject will receive his second month's study medication and medication/voiding and pain diaries.
2. Month Visit (Visit 3):

   Same as 1 Month Visit.
3. Month Visit (Visit 4):

First, the subject will be asked to fill out follow-up questionnaires

Next, the patient's caregiver will perform a physical exam and prostate massage during which, expressed prostatic secretions will be collected.

Then, his previous month's empty medication container and completed diaries will be collected. A pill count will then be done.

Finally, the subject will be sent to the Male Fertility Lab to collect a semen sample (as in Screening Visit).

12 Month Visit (Visit 5): With the exception of pill count, etc., same as Visit 3.

Dose:

* Active drug: Viagra, 50mg, orally, once a day, for 90 days
* Placebo: identically-appearing pill supplied by Pfizer

Concurrent Therapy:

_ No concurrent therapy will be offered

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of male Chronic Pelvic Pain Syndrome Type III
* Age 18 - 65
* Pelvic pain duration of at least 3 months

Exclusion Criteria:

* Urinary tract infection within the last year
* Sexually transmitted disease within 3 months
* Antiviral therapy or antibiotics within the last 3 months
* Currently taking any medications or recreational drugs containing nitrates 3A4 inhibitors such as erythromycin, ketoconazole, or itraconazole
* Alpha-blocker therapy for treatment of high blood pressure or prostate problems
* Suffered a heart attack, stroke or life-threatening arrhythmia within the last months
* Cardiac failure or coronary artery disease causing unstable angina
* Resting hypotension (BP<90/50) or hypertension (BP>170/110)
* Patients with retinitis pigmentosa
* Kidney, liver or blood problems (including sickle cell anemia or leukemia)
* Allergy to sildenafil
* Deformed penis, Peyronie's disease or ever having had an erection lasting more than 4 hours
* Stomach ulcers or any types of bleeding problems
* Use of any other medical treatments that cause erections: pills, medicines that are injected or inserted into the penis, implants or vacuum pumps
* Back pain, unilateral testicular pain or rectal pain only
* Post-surgical pain
* Prostate biopsy or cystoscopy within 3 months
* Pain from another source in the genital tract, such as kidney stones or neoplasm
* History of prostate, bladder, renal or other urinary malignancies
* History of intravesical Bacillus Calmette-Guerin (BCG)
* Ulcerative colitis or Crohn's disease
* Radiation therapy to pelvis
* History of genitourinary tuberculosis
* Any neurological abnormalities including spinal cord injury and stroke
* Overtly psychotic or suicidal
* Unable to understand the protocol

In addition, subjects will be asked to refrain from having any new treatment for prostatitis during the study period, but will be allowed to remain on stable chronic therapy that they have been receiving for 3 or more months

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-07; Study Completion 2007-07

PRIMARY OUTCOMES:
NIH-CPSI -pain scores at 3 and 12 month post tx follow-up
AUA Score - at 3 and 12 month post tx follow-up

SECONDARY OUTCOMES:
Graded Chronic Pain Scale (GCPS)-3 & 12 mo post tx f/u

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Berger, MD, Principal Investigator — Professor of Urology
Locations (1):
- University of Washington, Urology Clinic, Seattle, Washington, United States